CLINICAL TRIAL: NCT06327061
Title: A Social Diffusion Fatal Overdose Prevention Intervention: Assessing the Effectiveness of People Who Use Opioids as Peer Educators in Training Using & Non-using Networks on Overdose & Stigma Reduction
Brief Title: Social Network Overdose Prevention and Education Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA058659 (NIH); IRB00026607 (Other: JHSPH IRB)
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Drug Overdose
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Intervention Model Description: a standard two-group clinical trial, one group is the experimental, the other the control
Who Masked: Participant
Masking Description: Both groups receive overdose prevention training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Peer education and network support (Experimental): During sessions 1 and 2, participants will be taught information and skills pertaining to overdose prevention and response. During the 3rd session, participants will trained to talk to their non drug using network members in overdose prevention and response.
  Interventions: Behavioral: Network overdose prevention
- comparison: Standard of care of health education (Active Comparator): In one session, participants will receive the standard of care for overdose prevention.
  Interventions: Behavioral: Standard of care health education

INTERVENTIONS:
Behavioral: Network overdose prevention — Participants are taught overdose prevention methods with network members.
  Arms: Experimental: Peer education and network support
Behavioral: Standard of care health education — Participants will receive the standard of care for overdose prevention.
  Arms: comparison: Standard of care of health education

SUMMARY:
The purpose of this study is to test a social intervention focused on overdose prevention and care. In the investigators prior work, the investigators have shown that people who use opioids (PWUO) can be effective peer educators (PEs).

DETAILED DESCRIPTION:
The purpose of this study is to test a social intervention focused on overdose prevention and care. In the investigators prior work, the investigators have shown that people who use opioids (PWUO) can be effective peer educators (PEs). The investigators have utilized PEs for overdose prevention in interventions that have focused on training network members who use drugs to respond to an overdose. Yet, many overdoses are witnessed by people who do not use drugs. Additionally, many PWUO report using drugs at home and living with someone who does not use drugs, which highlights the importance of training non-using network members on overdose response. Based on pilot data, the investigators propose expanding an overdose peer education intervention to focus on non-using network members. The intervention seeks to prepare network members to respond to an overdose and normalize discussions about overdose prevention planning between index PWUO and non-using network members. The intervention condition consists of 3 individual sessions focused on overdose prevention and response. This condition is designed to train index study participants to be Peer Educators. In addition to the three sessions, the non-drug using network member will be offered one session. The control condition is only 1 session focused on overdose prevention and response. Both intervention and control participants will invite social network members to take part in data collection activities

ELIGIBILITY:
Inclusion Criteria:

* self-reported illicit opioid use at least 2 times in the past two weeks;
* age 18 and older;
* living in the Baltimore metropolitan region;
* willing to engage in peer education; and
* having and willing to recruit at least one non-using network member.

Exclusion Criteria:

Participants without the cognitive ability to provide informed consent and have the physical ability to participate in in-person intervention sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-29 (Estimated)

PRIMARY OUTCOMES:
Number of drug overdoses | 3-months
  Number of drug overdoses in prior three months
Participant drug use | 3-months
  Proportion of times participants tested positive for drugs of fentanyl and xylazine using test strips in the prior 3 months.

SECONDARY OUTCOMES:
Number of Network member contacts | 3-months
  Number of network members talked to about overdose prevention in prior 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States